CLINICAL TRIAL: NCT04217122
Title: Effect of Strawberry Consumption on the Microbiome in Healthy Subjects: A Pilot Study
Brief Title: Effect of Strawberry Consumption on the Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB#18-000312
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Microbiome
Keywords: Strawberry; polyphenols; cholesterol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strawberry intervention group (Experimental): Participants consume two packages of 13 g of standard strawberry powder in the morning and afternoon/evening per day for 4 weeks
  Interventions: Other: strawberry powder
- Placebo group (Placebo Comparator): Participants consume two packages of 13 grams placebo powder in the morning and afternoon/evening for 4 weeks.
  Interventions: Other: placebo powder

INTERVENTIONS:
Other: strawberry powder — Participants consume 2 packages of standard strawberry powder (13 g x 2) daily for 4 weeks
  Arms: Strawberry intervention group
Other: placebo powder — Participants consume 2 packages of placebo powder (13 g x 2) daily for 4 weeks
  Arms: Placebo group

SUMMARY:
This pilot study will assess the ability of daily consumption of two servings of California strawberries to alter gut microbiome composition, leading to increased bile secretion and decreased plasma cholesterol in a free-living population.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded, placebo controlled, parallel design. Thirty subjects will be randomized to consume two servings of standardized freeze-dried strawberry powder (2 x 13g) daily or placebo for 4 weeks, followed by 2 weeks of follow up with beige diet only to observe whether the effect can be sustained for 2 weeks. Blood will be collected at baseline (week 0), weeks 4 and week 6 after strawberry consumption. On the day prior to the study visits participants will collect a stool and a 24-hr urine sample and bring to the lab. In addition, body weight and composition will be determined and questionnaires and 3-day food record will be completed. Twenty-four hour urine content of pelargonidin glucuronide will be measured for compliance. Plasma and fecal cholesterol and bile acids will be determined at baseline (week 0) and weeks 4 and 6.

Subjects will be assigned an enrollment number after signing the informed consent form approved by the UCLA Medical Internal Review Board. Subjects will undergo a physical exam, complete medical history, and blood draw. A standard chem. panel will be performed at the UCLA clinical laboratory. Eligible subjects will be enrolled into the study upon completion of screening evaluations and will be randomized to the strawberry or placebo arm at their baseline visit.

The study will be conducted in healthy free-living subjects (18-55 years). Subjects consume 13 grams standard strawberry powder in the morning and afternoon/evening or placebo powder for 4 weeks. Subjects will be instructed to eat a beige diet (low fiber<10g and low polyphenols <3 servings of polyphenol rich fruit/vegetables per day) during the entire study period. 24 hr urine pelargonidin glucuronide will be measured at weeks 2 (baseline), 6 and 8 for compliance. In addition, pelargondin, ellagic acid, dimethylellagic acid glucuronide and urolithin glucuronide will be measured in plasma and urine to determine strawberry phytochemical bioavailability and intestinal/microbiome metabolic capacity. Participants will meet with the dietitian for assessment of habitual dietary pattern and instructions on maintain on a beige diet. A list of foods with high fiber and phenolic compounds will be provided and subjects are instructed to follow the diet during the entirety of the study.

A standardized freeze-dried strawberry powder and a strawberry placebo powder provided by the California Strawberry Commission will be used. Ten grams of freeze dried powder is equivalent to about 110 g fresh fruit. One serving of fresh strawberry (one cup) is estimated to weigh 144 g and therefore is equivalent to 13 g of freeze dried powder. Subjects will consume two packages of 13 g of strawberry powder per day. The powder can be mixed into beverages and consumed with breakfast and dinner.

Strawberry powder ingredients include Individually Quick Frozen (IQF) strawberries. Placebo powder ingredients include fructose, sucrose, dextrose, tapioca maltodextrin, modified food starch, erythritol, cellulose gum, citric acid (anhydrous), N-C Strawberry Flavor Natual WONF, xanthan gum, malic acid, sugar beet fiber, silicon dioxide, nat. strawberry-type flavor, FD&C Red #40, FD&C Yellow 6, FD&C Blue 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adults age 18-55 years old (females have to be premenopausal)
* Typically consume low fiber/polyphenol diet (beige diet)

Exclusion Criteria:

* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement which interfere with the absorption of polyphenols.
* History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
* Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Is known HIV positive (subjects who are HIV positive are known to have high evels of LDL cholesterol and generalized heart inflammation).
* Is unable or unwilling to comply with the study protocol.
* Using prebiotics, probiotics, yogurt, and/or any fiber supplements regularly
* Allergy or sensitivity to strawberries. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive affirmation by the subject of strawberry ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded.
* Taking antibiotics or laxatives within the past 3 months
* Any subject who demonstrate a risk of non-compliance with study procedure, or one who cannot read, understand or complete study - related materials in the opinion of the study investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change in microbiome composition | 4 weeks
  Change in phyla, genes and species of gut bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No